CLINICAL TRIAL: NCT00275886
Title: Activation and Recruitment of Gastric Infiltrating Lymphocytes During H. Pylori Infection
Brief Title: Activation and Recruitment of GIL During Hp Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701221
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 2005-12

CONDITIONS: Helicobacter Gastritis; Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Helicobacter pylori is a major human pathogen that infects over half of the world population. Infection initiates a series of changes in the gastric mucosa, beginning with gastritis and leading in some patients to peptic ulcer disease, mucosa-associated lymphomas, and gastric adenocarcinoma. It is believed that host factors, in particular, the T cell-mediated immune responses may play an important role in the pathogenesis of diseases induced by H. pylori infection. Recent results revealed that there were higher IFN-γ secreting cells in gastric infiltrating T cells isolated from H. pylori infected patients than in uninfected patients, suggesting that the TH1 response and degree of IFN-γ production is associated with disease severity. Meanwhile, recent studies have shown that apoptosis of the gastric epithelium is increased during infection and this response is associated with an expansion of gastric T-helper type 1 (Th1) cells. In this project, we are trying to further investigate role of host T cell mediated immune response in pathogenesis of Helicobacter infection by characterization of the expression of chemokine receptors on gastric infiltrating lymphocytes. We are going to investigate the mechanisms involving in chemokine/chemokine receptor interaction in recruitment of gastric infiltrating lymphocytes and pathogenesis of gastric mucosa damage in Helicobacter infection. This study will be helpful for understanding the mechanisms of activation and recruitment of gastric-infiltrating lymphocytes during gastric inflammation.

DETAILED DESCRIPTION:
Specific Aim #1: Characterization of the gastric infiltrating T cells from H. pylori gastritis patients A. Patients H. pylori infected gastritis and asymptomatic patients are selected from National Taiwan University hospital. The gastric biopsy specimen are taken from endoscopic biopsy in routine health check up or panendoscopic examination for the despeptic patients. HP negative gastritis patients will also be studied for negative control.

B. Immunohistochemical identification of T cells and expression of chemokine receptors.

Specific Aim #2 . Isolation and characterization of chemokines and chemokine receptors of the infiltrating lymphocytes in H. pylori-associated gastritis tissue

A. Isolation of gastric infiltrating lymphocyte B. Identification of the expression of chemokine receptor in gastric infiltrating lymphocytes by flow cytometry C. Detection of expression of chemokines in gastric tissues

ELIGIBILITY:
Inclusion Criteria:

* patients receiveing endoscopy examination due to dyspepsia

Exclusion Criteria:

* nil

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-01; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ning Hsu, MD, PhD, Principal Investigator — Department of Immunology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan